CLINICAL TRIAL: NCT04313530
Title: Study on the Effect and Mechanism of Transcranial Magnetic Stimulation in Multiple System Atrophy Patients With Fatigue
Brief Title: TMS Treatment in Multiple System Atrophy With Fatigue
Acronym: TMSMSAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Piu Chan, Director, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1225435380@qq.com
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Transcranial Magnetic Stimulation; Multiple System Atrophy; Fatigue
Keywords: TMS,MSA,fMRI,Fatigue,functional, connectivity
MeSH Terms: conditions — Multiple System Atrophy; Fatigue | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fatigue in MSA Arm one (Experimental): This arm will receive a total 10 sessions of TMS stimulation in two weeks. Pre and post intervention scales will be performed on week one, week 2 and week 4.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- fatigue in MSA Arm two (Sham Comparator): This arm will receive a total 10 sessions of sham-TMS stimulation in two weeks. Pre and post intervention scales will be performed on week one, week 2 and week 4.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a non-invasive method that uses electromagnetic induction to produce electric currents in the cortex that are strong enough to depolarise neurons sufficiently to trigger action potentials. It is an outpatient based procedure that when used in conjunction with a neuro-navigation system, specific cortical areas can be targeted for greater accuracy and efficacy. In clinical studies, TMS is delivered as trains of pulses (repetitive TMS, rTMS) to prolong its effects. While the exact mechanism of TMS treatment fatigue is unknown, it is thought to regulate the activity of the complex cortical and subcortical networks connectivity changes involved in the processing of fatigue signals.

SUMMARY:
Transcranial magnetic stimulation (TMS) is a procedure that has been shown to improve fatigue in chronic sufferers. It uses a plastic covered coil that sends a magnetic pulse through the skull into the brain and by targeting particular areas in the brain it can be used to help modulate the perception of fatigue.

The study intends to use this technique to treat such a disabling symptom in patients who suffer from Multiple System Atrophy (MSA). Initially the aim is to study this technique in 22 MSA patients who are suffering from fatigue . These patients would require an resting-state funtional MRI before and after the stimulation. The stimulation would be performed ten sessions and the patients would be assessed by a clinician using well recognized clinical tools.

It is anticipated that there will be a meaningful improvement in fatigue. It is also anticipated that TMS is a safety technique to use in MSA patients . Our findings will revealed that fatigue may be associated with an altered default mode network and sensorimotor network connectivity in MSA patients. We hypothesize that these divergent motor and cognitive networks connectivity changes and their adaptive or maladaptive functional outcome may play a prominent role in the pathophysiology of fatigue in MSA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Multiple system atrophy diagnosed as "possible" or "probable" according to the 2008 MDS clinical diagnostic criteria;
2. Age ≥30Aged ≤ 75years old;
3. right handedness
4. MMSE>24
5. the dosage and species of anti-parkinson drug is maintained during the treatment;
6. The patient or his/her legal guardian agreed to participate in the trial and signed the informed consent.Ability to follow research plans and visit plans.
7. FSS≥4

Exclusion Criteria:

1. Serious medical and mental illness;
2. History of stroke, intracranial tumor and other central nervous system;
3. Patients with suicidal tendencies and psychotic symptoms.
4. MRI for contraindications, such as metal implants, claustrophobia, etc
5. Contraindications for TMS (such as history of seizures, pregnant women, installation of pacemakers, metal inclusions in the body, intracranial hypertension, severe bleeding tendency, etc.)
6. Patients who received TMS treatment for nearly half a year.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Fatigue Severity Scale-9 (FSS-9) | Pre-treatment, post-treatment 0, 2, 4 weeks
  To quantify changes of the severity of fatigue.The higher the score, the worse the fatigue.

SECONDARY OUTCOMES:
Changes in 17-item Hamilton Depression Scale(HAMD-17) | Pre-treatment, post-treatment 0, 2, 4 weeks
  To quantify changes of the severity of depression.The higher the score, the worse the depression.
Changes in Hamilton Anxiety Scale(HAMA) | Pre-treatment, post-treatment 0, 2, 4 weeks
  To quantify changes of the severity of anxiety.The higher the score, the worse the anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Biao Chen, MD,PHD, Study Chair — Xuanwu Hospital of Capital Medical University
Locations (1):
- The Neurology Department of Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China